CLINICAL TRIAL: NCT04382118
Title: Var_DFO:Open Versus Closed Wedge Distal Femoral Varus Osteotomy for the Valgus Knee. Indications, Clinical and Radiological Outcome
Brief Title: Open Versus Closed Wedge Distal Femoral Varus Osteotomy for the Valgus Knee. Indications, Clinical and Radiological Outcome
Acronym: Var_DFO
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00108; ch20Muendermann3
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Valgus Malalignment of the Knee
Keywords: Closed Wedge Distal Femoral Varus Osteotomy (CWDFO); Open Wedge Distal Femoral Varus Osteotomy (OWDFO)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OWDFO: Open Wedge Distal Femoral Varus osteotomy
  Interventions: Other: Data collection from routine medical records
- CWDFO: Closed Wedge Distal Femoral Varus osteotomy
  Interventions: Other: Data collection from routine medical records

INTERVENTIONS:
Other: Data collection from routine medical records — Data collection from routine medical records (clinical and radiological data)

SUMMARY:
This study is to analyze the indications of the two most popular techniques of distal femoral osteotomy (DFO) performed in patients with valgus malalignment and symptomatic degenerative changes in the lateral compartment of the knee and to evaluate the clinical and radiological outcome of a case series of patients who have received this operation at the Department of Orthopaedics and Traumatology and the Department of Surgery of the University Hospital Basel.

ELIGIBILITY:
Inclusion Criteria:

* patients who received a distal femoral osteotomy (DFO) for valgus knee osteoarthritis between 1.1.2013 and 31.12.2017

Exclusion Criteria:

* Absence of informed consent
* Absence of X-Rays documenting the preoperative deformity or postoperative result

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received a DFO for valgus knee arthritis at the Clinic of Orthopaedics and Traumatology at the University Hospital Basel between 1.1.2013 and 31.12.2017 will be included in this study.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of the correction of the deformity | at Baseline
  The mechanical axis of the femur and the tibia and hence the mechanical tibiofemoral angle (MFTA) will be measured pre- and postoperatively. (the goal of the operation is a neutral alignment, MFTA angle of 0°)

SECONDARY OUTCOMES:
incidence of disruptive hardware | at Baseline
  Information regarding the incidence of disruptive hardware and of hardware removal operations because of this, time needed until bony union is achieved, complications, delayed and non-union rates and need of conversion to arthroplasty
pain level | at Baseline
  Information regarding pain levels measured with visual analog scale score (VAS). The visual analogue scale (VAS) is a scale used to determine the pain intensity experienced by individuals. It consists of a line, approximately 10-15 cm in length, with the left side signifying no pain with a smiling face image and the right side signifying the worst pain.
pain medication intake preoperatively and at the final follow up | at Baseline
  pain medication intake preoperatively and at the final follow up

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Muendermann, Prof. Dr. med., Principal Investigator — Department of Orthopaedics and Traumatology, University Hospital Basel
Locations (1):
- Clinic for Orthopaedics and Traumatology, University Hospital basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Ismailidis P, Schmid C, Werner J, Nuesch C, Mundermann A, Pagenstert G, Egloff C. Distal femoral osteotomy for the valgus knee: indications, complications, clinical and radiological outcome. Arch Orthop Trauma Surg. 2023 Oct;143(10):6147-6157. doi: 10.1007/s00402-023-04923-w. Epub 2023 Jun 6. PMID 37278744